CLINICAL TRIAL: NCT00098735
Title: Efficacy and Safety of FTY720 in Patients Who Receive a Kidney Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720A2302
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Kidney Transplantation
Keywords: Kidney,Transplantation, rejection, immunosuppression
MeSH Terms: conditions — Rejection, Psychology | interventions — Fingolimod Hydrochloride

INTERVENTIONS:
Drug: FTY720

SUMMARY:
In patients who receive an organ transplant, their body considers this organ as foreign and attempts to destroy it. This is called rejection. All patients who receive an organ transplant, will take a combination of anti-rejection medications. These medications prevent the new organ from being rejected from the body. FTY720 is a new compound that helps prevent organ rejection.

ELIGIBILITY:
Inclusion Criteria:

* First kidney transplantation
* Male and female patients
* Between 18 and 65 years old

Exclusion Criteria:

* Patient in need of multi-organ transplant
* Patients with history of cardiac arrest
* Patients with any past or present malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2004-04; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
IA, IB, IIA, IIB, III, or humoral rejection diagnosed by biopsy according to Banff 97 criteria within 6 months post transplant
Permanent resumption of dialysis within 6 months post transplant
Surgical removal of graft within 6 months post transplant
Death within 6 months post transplant
Withdrawal of consent, death, or lost to follow up within 6 months post transplant

SECONDARY OUTCOMES:
IA, IB, IIA, IIB, III, or humoral rejection diagnosed by biopsy according to Banff 97 criteria within 12 months post transplant
Permanent resumption of dialysis within 12 months post transplant
Surgical removal of graft within 12 months post transplant
Death within 12 months post transplant
Withdrawal of consent, death, or lost to follow up within 12 months post transplant
Serum creatinine, estimated creatinine clearance, abnormalities of vital signs and laboratory variables and measurements of urine protein at Days 0, 1, 7, 14 and 28, Months 3, 6, 9 and 12.
FEV1 , FVC, FEV1/FVC, DLCO and FEF 25%-75% at Day 28, Months 6 and 12
Absolute lymphocyte count at Days 0, 1, 7, 14 and 28, Months 3, 6, 9 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: NOVARTIS, Study Director — Novartis

REFERENCES:
- [Result] Tedesco-Silva H, Mourad G, Kahan BD, Boira JG, Weimar W, Mulgaonkar S, Nashan B, Madsen S, Charpentier B, Pellet P, Vanrenterghem Y. FTY720, a novel immunomodulator: efficacy and safety results from the first phase 2A study in de novo renal transplantation. Transplantation. 2005 Jun 15;79(11):1553-60. PMID 15940045